CLINICAL TRIAL: NCT01874288
Title: A Phase I/II Study of De-immunized DI-Leu16-IL2 Immunocytokine Administered Subcutaneously in Patients With B-cell Non-Hodgkin Lymphoma (NHL)
Brief Title: A Study of De-immunized DI-Leu16-IL2 Administered Subcutaneously in Participants With B-cell NHL
Acronym: DI-Leu16-IL2
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Clinical benefit was noted in the earlier portion of the trial; hence, participants were not enrolled in 2 expansion cohorts and the study was terminated early.
Sponsor: Alopexx Oncology, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AO-101
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: B-cell Non-Hodgkin Lymphoma
Keywords: NHL; Immunocytokine; Lymphoma; Non-Hodgkin; B-cell; IL (interleukin)
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- DI-Leu16-IL2 0.5 mg/m^2 (Experimental): Participants will receive DI-Leu16-IL2 0.5 mg/m^2 subcutaneously (SC) for 3 consecutive days every 3 weeks (21-day cycle) for a total of 4 cycles.
  Interventions: Drug: DI-Leu16-IL2
- DI-Leu16-IL2 1.0 mg/m^2 (Experimental): Participants will receive DI-Leu16-IL2 1.0 mg/m^2 SC for 3 consecutive days every 3 weeks (21-day cycle) for a total of 4 cycles.
  Interventions: Drug: DI-Leu16-IL2
- DI-Leu16-IL2 2.0 mg/m^2 (Experimental): Participants will receive DI-Leu16-IL2 2.0 mg/m^2 SC for 3 consecutive days every 3 weeks (21-day cycle) for a total of 4 cycles.
  Interventions: Drug: DI-Leu16-IL2
- DI-Leu16-IL2 4.0 mg/m^2 (Experimental): Participants will receive DI-Leu16-IL2 4.0 mg/m^2 SC for 3 consecutive days every 3 weeks (21-day cycle) for a total of 4 cycles
  Interventions: Drug: DI-Leu16-IL2
- DI-Leu16-IL2 6.0 mg/m^2 (Experimental): Participants will receive DI-Leu16-IL2 6.0 mg/m^2 SC for 3 consecutive days every 3 weeks (21-day cycle) for a total of 4 cycles.
  Interventions: Drug: DI-Leu16-IL2

INTERVENTIONS:
Drug: DI-Leu16-IL2 — DI-Leu16-IL2 will be administered per dose and schedule specified in the arm.

SUMMARY:
This dose-escalation study is designed for determining the safety, tolerability, pharmacokinetics (PK), biological, and clinical activity of DI-Leu16-IL2 administered to participants with cluster of differentiation 20 (CD20) positive NHL that have failed standard rituximab-containing therapy.

DETAILED DESCRIPTION:
The participants will be enrolled during dose escalation and during 2 expansion cohorts of up to 12 participants each.

The dose escalation portion of the trial will incorporate a modified accelerated titration design. Therefore, the trial will enroll 3 participants per dose level with a doubling of the dose at each level during the accelerated stage of the study (skipping every other dose level). Once the first instance of any Grade 3 or higher treatment related toxicity (with some notable exceptions) is observed on the first cycle, the accelerated stage will end and the trial will revert to a conventional design using cohorts of 3 or 6 participants (standard 3+3 design), with single step 2 milligrams (mg)/square meter (m^2) increments.

To further explore the clinical efficacy, additional participants (up to 12 per cohort) may be enrolled at the optimal biologic dose (OBD) or maximum tolerated dose (MTD).

At the end of the study, participants may be enrolled into an open-label extension study (AO-101-EXT [NCT02151903]), at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with CD20-expressing B-cell NHL that is relapsed or refractory to standard therapy. Chronic lymphocytic leukemia/small lymphocytic lymphoma with peripheral blood leukemia/lymphoma cells and high-grade lymphomas are excluded.
2. Participants must have received prior rituximab-containing therapy.
3. Evaluable disease. In the absence of lymphadenopathy, splenomegaly with defects or measurable extra-medullary disease is acceptable.
4. Participants who have received a prior autologous stem cell transplant are eligible if the transplant occurred >6 months ago.
5. Participants who have received a prior allogeneic stem cell transplant are eligible if:

   1. The transplant occurred >6 months ago
   2. There is no evidence of active graft versus host disease
   3. Systemic immunosuppressive agents (including corticosteroids) have not been received for at least 8 weeks
6. Karnofsky performance scale ≥70%
7. Life expectancy ≥12 weeks
8. Adequate baseline functions:

   1. Serum creatinine ≤1.5 mg/deciliter (dL)
   2. Total white blood cell (WBC) count ≥3000/microliter (µL) or absolute neutrophil count (ANC) ≥1000/µL
   3. Absolute lymphocyte count ≥0.75 * 10^3/µL
   4. Platelet count ≥75,000/µL
   5. Hematocrit ≥25% or hemoglobin ≥9 grams/100 milliliters (mL)
   6. Alanine aminotransferase (ALT) <2.5 * upper limit of normal (ULN)
   7. Aspartate aminotransferase (AST) <2.5 * ULN
   8. Total bilirubin (TBili) <1.5 * ULN
   9. Sodium, potassium, and phosphorus levels no worse than grade 1
   10. Chest x-ray (CXR) or computed tomography (CT) within 4 weeks prior to Day 1 with no evidence of pulmonary congestion, pleural effusions, pulmonary fibrosis, or significant emphysema. If results are questionable, participants should have additional lung function testing to exclude clinically relevant restriction or obstruction. Participants must have a forced expiratory volume (FEV-1) and diffusing capacity of the lung for carbon monoxide (DLCO) of at least 65% and 50% of expected, respectively.
   11. Electrocardiogram (12-lead ECG) QTc ≤480 millisecond (ms)
   12. Cardiac stress test (for example, stress thallium scan, stress echocardiography) with normal results if participant is suspected to have coronary artery disease.
9. Participants participating in the study are to use adequate birth control measures (abstinence, oral contraceptives, barrier method with spermicide or surgical sterilization) during the study. Females of childbearing potential must have a negative serum pregnancy test on the days of dosing. A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (that is, has had menses at any time in the preceding 24 consecutive months).
10. Provide written informed consent prior to any screening procedures

Exclusion Criteria:

1. Evidence of central nervous system lymphoma or lymphomatous meningitis
2. Prior treatment with interleukin 2 (IL2) within the last 5 years
3. Type I hypersensitivity or anaphylactic reactions to murine proteins or to previous infusion of rituximab
4. Pregnant or lactating female
5. An immediate need for palliative radiotherapy or systemic corticosteroid therapy
6. Known intercurrent infections (including hepatitis C virus and human immunodeficiency virus or other conditions), or clinical evidence of these conditions
7. Actively infected with or chronic carriers of hepatitis B virus as demonstrated by positive hepatitis B core antibody or hepatitis B surface antigen. Participants who are seropositive only, that is, surface antibody positive [HbsAb], are permitted.
8. Other significant active infection.
9. Major surgery, chemotherapy, investigational agent, or radiation within 30 days of Day 1
10. Uncontrolled hypertension (diastolic greater to or equal to 100 millimeters of mercury [mmHg]) or hypotension (systolic less than or equal to 90 mmHg)
11. History of repeated and clinically relevant episodes of syncope or other paroxysmal, ventricular, or other significant arrhythmias
12. History of medically significant ascites requiring repetitive paracentesis
13. Previous diagnosis of autoimmune disease (Exceptions: participants with autoimmune thyroiditis or vitiligo may be enrolled)
14. Organ transplant recipient
15. History of prior therapy or a serious, uncontrolled medical disorder that in the Investigator's opinion would impair participation in the study
16. Known hypersensitivity to Tween-80 or human immunoglobulin
17. Legal incapacity or limited legal capacity
18. Participants with bulky lymph nodes (LNs) (≥10 centimeters [cm]) or marked splenomegaly (that is, extending into pelvis or crossing the midline).
19. Circulating levels of rituximab >75.0 micrograms (µg)/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-11-25 (Actual); Primary Completion 2014-01-27 (Actual); Study Completion 2016-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Vlock, MD, Study Director — Alopexx Oncology, LLC
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - St. Jude Hospital Yorba Linda, Fullerton, California
  - University of Minnesota, Minneapolis, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Joe Arlington Cancer Research and Treatment Center, Lubbock, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] King DM, Albertini MR, Schalch H, Hank JA, Gan J, Surfus J, Mahvi D, Schiller JH, Warner T, Kim K, Eickhoff J, Kendra K, Reisfeld R, Gillies SD, Sondel P. Phase I clinical trial of the immunocytokine EMD 273063 in melanoma patients. J Clin Oncol. 2004 Nov 15;22(22):4463-73. doi: 10.1200/JCO.2004.11.035. Epub 2004 Oct 13. PMID 15483010
- [Background] Ko YJ, Bubley GJ, Weber R, Redfern C, Gold DP, Finke L, Kovar A, Dahl T, Gillies SD. Safety, pharmacokinetics, and biological pharmacodynamics of the immunocytokine EMD 273066 (huKS-IL2): results of a phase I trial in patients with prostate cancer. J Immunother. 2004 May-Jun;27(3):232-9. doi: 10.1097/00002371-200405000-00008. PMID 15076141
- [Background] Maloney DG, Liles TM, Czerwinski DK, Waldichuk C, Rosenberg J, Grillo-Lopez A, Levy R. Phase I clinical trial using escalating single-dose infusion of chimeric anti-CD20 monoclonal antibody (IDEC-C2B8) in patients with recurrent B-cell lymphoma. Blood. 1994 Oct 15;84(8):2457-66. PMID 7522629
- See also: Sponsor website — http://www.alopexx.com
- See also: National Cancer Institute at the National Institute of Health — http://www.cancer.gov/cancertopics/types/non-hodgkin

RESULTS

PARTICIPANT FLOW:
Groups:
- DI-Leu16-IL2 0.5 mg/m^2: Participants received DI-Leu16-IL2 0.5 milligrams per square meter (mg/m^2) subcutaneously (SC) for 3 consecutive days every 3 weeks (21-day cycle) for a total of 4 cycles.
- DI-Leu16-IL2 1.0 mg/m^2: Participants received DI-Leu16-IL2 1.0 mg/m^2 SC for 3 consecutive days every 3 weeks (21-day cycle) for a total of 4 cycles.
- DI-Leu16-IL2 2.0 mg/m^2: Participants received DI-Leu16-IL2 2.0 mg/m^2 SC for 3 consecutive days every 3 weeks (21-day cycle) for a total of 4 cycles.
- DI-Leu16-IL2 4.0 mg/m^2: Participants received DI-Leu16-IL2 4.0 mg/m^2 SC for 3 consecutive days every 3 weeks (21-day cycle) for a total of 4 cycles.
- DI-Leu16-IL2 6.0 mg/m^2: Participants received DI-Leu16-IL2 6.0 mg/m^2 SC for 3 consecutive days every 3 weeks (21-day cycle) for a total of 4 cycles.
Period: Overall Study
Arm/Group | DI-Leu16-IL2 0.5 mg/m^2 | DI-Leu16-IL2 1.0 mg/m^2 | DI-Leu16-IL2 2.0 mg/m^2 | DI-Leu16-IL2 4.0 mg/m^2 | DI-Leu16-IL2 6.0 mg/m^2
Started | 3 | 3 | 9 | 7 | 2
Received at Least 1 Dose of Study Drug | 3 | 3 | 9 | 7 | 2
Completed | 0 | 3 | 4 | 0 | 0
Not Completed | 3 | 0 | 5 | 7 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Progressive disease | 2 | 0 | 3 | 5 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Groups:
- DI-Leu16-IL2 0.5 mg/m^2: Participants received DI-Leu16-IL2 0.5 mg/m^2 SC for 3 consecutive days every 3 weeks (21-day cycle) for a total of 4 cycles.
- Total: Total of all reporting groups
Arm/Group | DI-Leu16-IL2 0.5 mg/m^2 | DI-Leu16-IL2 1.0 mg/m^2 | DI-Leu16-IL2 2.0 mg/m^2 | DI-Leu16-IL2 4.0 mg/m^2 | DI-Leu16-IL2 6.0 mg/m^2 | Total
Number analyzed (Participants) | 3 | 3 | 9 | 7 | 2 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (12.22) | 66.7 (14.84) | 64.0 (11.55) | 59.6 (9.61) | 57.5 (13.44) | 60.9 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 6 | 0 | 2 | 10
  Male | 2 | 2 | 3 | 7 | 0 | 14
Tumor Measurement: Sum of Product of Diameters [Mean (Standard Deviation); unit: centimeters (cm)] | 15.11667 (9.726296) | 12.21667 (12.110806) | 17.63953 (16.388997) | 27.95857 (22.005858) | 27.86500 (10.896515) | 20.50816 (16.836733)
Tumor Measurement: Sum of Longest of Diameters [Mean (Standard Deviation); unit: cm] | 6.000 (3.0414) | 6.133 (4.3524) | 9.462 (5.4068) | 11.100 (5.1901) | 10.300 (5.6569) | 9.161 (4.9829)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of DI-Leu16-IL2
Description: The MTD was determined based on toxicities from the first 2 cycles of treatment. The MTD was the highest dose tested with no more than 1 participant out of 6 experienced a dose-limiting toxicity (DLT). All non-hematologic adverse events (AEs) and all hematologic AEs of greater than Grade 3 were considered relevant to determining DLTs. DLTs included absolute lymphocyte count (ALC) Grade 3 and 4 (if ALC does not resolve to baseline grade according to Common Terminology Criteria for Adverse Events (CTCAE) v4 within 5 days post the final injection per cycle of DI-Leu16-IL2), and absolute neutrophil count (ANC) Grade 3 (If ANC does not resolve to at least Grade 2 within 5 days post the final injection per cycle of DI-Leu16-IL2) and Grade 4 (any).
Time Frame: First 2 cycles of treatment (each cycle = 21 days)
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: mg/m^2
Groups:
- DI-Leu16-IL2: Participants received assigned doses of DI-Leu16-IL2 SC for 3 consecutive days every 3 weeks (21-day cycle) for a total of 4 cycles.
Arm/Group | DI-Leu16-IL2
Number analyzed (Participants) | 24
mg/m^2 | 4.0

2. Primary Outcome: Number of Participants With a DLT
Description: All non-hematologic AEs and all hematologic AEs of greater than Grade 3 were considered relevant to determining DLTs. DLTs included ALC Grade 3 and 4 (if ALC does not resolve to baseline grade according to CTCAE v4 within 5 days post the final injection per cycle of DI-Leu16-IL2), and ANC Grade 3 (If ANC does not resolve to at least Grade 2 within 5 days post the final injection per cycle of DI-Leu16-IL2) and Grade 4 (any).
Time Frame: First 2 cycles of treatment (each cycle = 21 days)
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | DI-Leu16-IL2 0.5 mg/m^2 | DI-Leu16-IL2 1.0 mg/m^2 | DI-Leu16-IL2 2.0 mg/m^2 | DI-Leu16-IL2 4.0 mg/m^2 | DI-Leu16-IL2 6.0 mg/m^2
Number analyzed (Participants) | 3 | 3 | 9 | 7 | 2
Participants | 0 | 0 | 0 | 0 | 2

3. Primary Outcome: Number of Participants With Best Overall Response (BOR) Assessed Per International Workshop for Non-Hodgkin Lymphoma (NHL) Response Criteria
Description: BOR included complete response (CR), unconfirmed CR (CRu), partial response (PR), stable disease (SD), and progressive disease (PD). CR: 1) Disappearance of all detectable clinical and radiological evidence of disease; 2) lymph nodes (LN) regressed to normal size; 3) other organs (spleen, liver, kidneys) that were enlarged before therapy must have decreased in size; 4) clear bone marrow (BM) infiltrate. CRu: must meet CR criteria 1 and 3, as well as ≥1 of following: residual LN mass >1.5 cm in greatest transverse diameter; individual nodes that were previously confluent regressed by >75% in sum of product diameters (SPD); or indeterminate BM. PR: 6 largest dominant nodes or nodal masses decreased by ≤50% in SPD; no increase in size of other nodes; liver or spleen; splenic and hepatic nodules regressed ≥50% in SPD; and no new disease. SD: less than a PR but not PD. PD: 50% increase from nadir in SPD of any abnormal node for PR or nonresponders and appearance of any new lesion.
Time Frame: First dose of study drug until first appearance of CR, CRu, PR, SD, or PD (up to 6 months)
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | DI-Leu16-IL2 0.5 mg/m^2 | DI-Leu16-IL2 1.0 mg/m^2 | DI-Leu16-IL2 2.0 mg/m^2 | DI-Leu16-IL2 4.0 mg/m^2 | DI-Leu16-IL2 6.0 mg/m^2
Number analyzed (Participants) | 3 | 3 | 9 | 7 | 2
Participants
  CR | 0 | 0 | 2 | 1 | 0
  CRu | 0 | 0 | 0 | 0 | 0
  PR | 0 | 1 | 1 | 0 | 0
  SD | 2 | 2 | 1 | 2 | 0
  PD | 1 | 0 | 4 | 4 | 2

4. Primary Outcome: Tumor Measurement: Percent Change From Baseline in Sum of Product of Diameters at the End of Study
Description: Sum of product diameters sums the product of the 2 tumor measurements on each lesion. If only 1 measurement was available, it was used as the longest length and the product of the lengths in the sum. Baseline value is the last non-missing measurement prior to receiving study drug injection. None of the participants were considered evaluable in 'DI-Leu16-IL2 0.5 mg/m^2' arm for this outcome measure at the end of study, and therefore, data were not collected for that arm.
Time Frame: Baseline, end of study (EOS) (up to approximately 3 years)
Population: Safety population included all enrolled participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | DI-Leu16-IL2 0.5 mg/m^2 | DI-Leu16-IL2 1.0 mg/m^2 | DI-Leu16-IL2 2.0 mg/m^2 | DI-Leu16-IL2 4.0 mg/m^2 | DI-Leu16-IL2 6.0 mg/m^2
Number analyzed (Participants) | 0 | 3 | 5 | 5 | 2
percent change |  | -31.54881 (60.445273) | -26.37248 (78.719865) | 48.83017 (120.291120) | 87.98408 (78.864919)

5. Primary Outcome: Tumor Measurement: Percent Change From Baseline in Sum of Longest Diameters at the End of Study
Description: Sum of longest diameters is the sum of the longest measured length of each tumor lesion. Baseline value is the last non-missing measurement prior to receiving study drug injection. None of the participants were considered evaluable in 'DI-Leu16-IL2 0.5 mg/m^2' arm for this outcome measure at the end of study, and therefore, data were not collected for that arm.
Time Frame: Baseline, EOS (up to approximately 3 years)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | DI-Leu16-IL2 0.5 mg/m^2 | DI-Leu16-IL2 1.0 mg/m^2 | DI-Leu16-IL2 2.0 mg/m^2 | DI-Leu16-IL2 4.0 mg/m^2 | DI-Leu16-IL2 6.0 mg/m^2
Number analyzed (Participants) | 0 | 3 | 5 | 5 | 2
percent change |  | -30.657 (60.3132) | -27.412 (49.2553) | 1.398 (43.4731) | 28.516 (22.5263)

6. Secondary Outcome: Number of Participants With Anti-DI-Leu16-IL2 Antibodies
Time Frame: First dose of study drug up to EOS (up to approximately 3 years)
Population: Due to early termination of study, data for this outcome measure were not collected.
Arm/Group | DI-Leu16-IL2 0.5 mg/m^2 | DI-Leu16-IL2 1.0 mg/m^2 | DI-Leu16-IL2 2.0 mg/m^2 | DI-Leu16-IL2 4.0 mg/m^2 | DI-Leu16-IL2 6.0 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug up to EOS (up to approximately 3 years)
Description: Safety population included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | DI-Leu16-IL2 0.5 mg/m^2 | DI-Leu16-IL2 1.0 mg/m^2 | DI-Leu16-IL2 2.0 mg/m^2 | DI-Leu16-IL2 4.0 mg/m^2 | DI-Leu16-IL2 6.0 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/9 | 0/7 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/3 | 1/9 | 3/7 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 9/9 | 7/7 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DI-Leu16-IL2 0.5 mg/m^2 (N=3) | DI-Leu16-IL2 1.0 mg/m^2 (N=3) | DI-Leu16-IL2 2.0 mg/m^2 (N=9) | DI-Leu16-IL2 4.0 mg/m^2 (N=7) | DI-Leu16-IL2 6.0 mg/m^2 (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DI-Leu16-IL2 0.5 mg/m^2 (N=3) | DI-Leu16-IL2 1.0 mg/m^2 (N=3) | DI-Leu16-IL2 2.0 mg/m^2 (N=9) | DI-Leu16-IL2 4.0 mg/m^2 (N=7) | DI-Leu16-IL2 6.0 mg/m^2 (N=2)
Injection site erythema (General disorders) | 2 | 3 | 7 | 6 | 2
Injection site pruritus (General disorders) | 3 | 3 | 6 | 4 | 1
Chills (General disorders) | 1 | 1 | 5 | 7 | 2
Fatigue (General disorders) | 1 | 3 | 4 | 6 | 1
Pyrexia (General disorders) | 1 | 1 | 5 | 3 | 2
Injection site induration (General disorders) | 1 | 2 | 4 | 3 | 0
Injection site rash (General disorders) | 1 | 1 | 3 | 4 | 1
Pain (General disorders) | 0 | 3 | 2 | 3 | 1
Injection site pain (General disorders) | 1 | 2 | 2 | 1 | 1
Oedema peripheral (General disorders) | 0 | 2 | 2 | 1 | 1
Injection site oedema (General disorders) | 0 | 1 | 3 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 5 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 4 | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 3 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 6 | 5 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 1 | 2
Lymphocyte count decreased (Investigations) | 0 | 0 | 4 | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 1 | 2
Platelet count decreased (Investigations) | 0 | 0 | 3 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 5 | 3 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 4 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 2 | 2
Hypotension (Vascular disorders) | 0 | 1 | 2 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 2 | 2 | 0
Injection site swelling (General disorders) | 1 | 1 | 1 | 1 | 0
Injection site discolouration (General disorders) | 0 | 0 | 3 | 0 | 0
Injection site inflammation (General disorders) | 1 | 0 | 2 | 0 | 0
Injection site warmth (General disorders) | 1 | 2 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 2 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Feeling cold (General disorders) | 1 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Infusion site haematoma (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site anaesthesia (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site discomfort (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site dryness (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site mass (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site nodule (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site vesicles (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Oral Pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 2 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 2 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 2 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT interval (Investigations) | 0 | 0 | 1 | 0 | 0
General physical condition abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0
Mean cell haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0
Protein total increased (Investigations) | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Central obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 2 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Sleep disorder due to general medical condition, insomnia Type (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 1 | 1 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Incision site pruritus (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Sinus operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Clinical benefit was noted in the earlier portion of the trial; hence, participants were not enrolled in 2 expansion cohorts and the study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less